CLINICAL TRIAL: NCT03141411
Title: Assisted Versus Manual Goal Directed Fluid Therapy in Major Abdominal Surgery
Brief Title: Assisted Fluid Management vs Manual GDFT
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2017/234 - B406201731981
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-04

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Goal-directed fluid therapy (GDFT) strategies based on cardiac output (CO) optimization have been shown to benefit moderate- to high-risk surgery patients and have recently been recommended by professional societies in the UK, in France, and in Europe. However, despite the growing evidence, these strategies are often not implemented in current practice. One of the reasons for this lack of implementation is that GDFT strategies, like any other complex clinical protocol, require significant provider attention and vigilance for consistent implementation and it is well known that even under study conditions protocol compliance rates are often not greater than 50%. To overpass this problem, our CO monitoring devices (EV1000, Edwards Lifesciences) have now an incorporated assisted fluid management software. This software determines fluid responsiveness by estimating the predicted change in stroke volume and suggests to the anesthesiologist when fluid is required .

DETAILED DESCRIPTION:
The aim of this study was to assess an assisted fluid management strategy in a moderate-to-high risk surgical cohort and compare that cohort to matched patients who received manual GDFT. Our hypothesis was that the assisted fluid management system would result in higher mean percentage time spent during surgery with a SVV < 13%

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing major abdominal surgery and requiring a CO monitoring for fluid management

Exclusion Criteria:

Emergency surgery Arrhythmia (e.g. atrial fibrillation) Aortic regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing major abdominal surgery and requiring a CO monitoring for fluid management
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
percentage time spent with SVV < 13% | intraoperative period
  defined as preload independent state

SECONDARY OUTCOMES:
amount of fluid administered | intraoperative period
  amount of cristalloid ( baseline ) AND fluid boluses (250 ml) received
amount of vasopressors required | intraoperative period
  amount of ephedrine, phenylephrine and norepinephrine
fluid balance | intraoperative period
  FLUID IN - FLUID OUT
incidence of major and minor complications | until 30 days post surgery
  see study protocol NCT03039946 for the description of these complications
PACU/ICU and hospital length of stay | until 30 days post surgery
  time spent in ICU and PACU

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, M.D, Principal Investigator — Erasme
Locations (1):
- Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Joosten A, Hafiane R, Pustetto M, Van Obbergh L, Quackels T, Buggenhout A, Vincent JL, Ickx B, Rinehart J. Practical impact of a decision support for goal-directed fluid therapy on protocol adherence: a clinical implementation study in patients undergoing major abdominal surgery. J Clin Monit Comput. 2019 Feb;33(1):15-24. doi: 10.1007/s10877-018-0156-x. Epub 2018 May 19. PMID 29779129